CLINICAL TRIAL: NCT03094000
Title: A Randomized Controlled Trial Examining Mindfulness Training Effect on Self-monitoring Adherence and Group Cognitive-behavioral Treatment Outcomes Among Women Suffering From Eating Disorders
Brief Title: Mindfulness Training Effect on Self-monitoring Adherence and Group CBT Outcomes for Binge Eating Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shalvata Mental Health Center (Other)
Collaborators: University of Haifa (Other); The Touro College and University System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHA-0019-13
Record Dates: First submitted 2017-02-19; First posted 2017-03-29 (Actual); Last update posted 2017-03-29 (Actual); Status verified 2017-03

CONDITIONS: Bulimia Nervosa; Binge-Eating Disorder; Night-eating Syndrome
Keywords: Bulimia Nervosa; Binge-Eating; Self monitoring; Cognitive Behavioral Therapy (CBT); Mindfulness
MeSH Terms: conditions — Bulimia Nervosa; Binge-Eating Disorder; Night Eating Syndrome

STUDY DESIGN:
Intervention Model Description: Following an evaluation and screening process, those who fit the criteria will be allocated randomly to one of the two research groups: experiment or control.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (CBTE-MIND) (Experimental): Adding a mindfulness skills intervention to group psychotherapy according to the principles of the Enhanced Cognitive-Behavioral Therapy (CBT-E) for eating disorders (Fairburn, 2008)
  Interventions: Behavioral: MIND; Behavioral: CBT-E
- Control group (CBTE) (Active Comparator): Group psychotherapy according to the principles of the Enhanced Cognitive-Behavioral Therapy (CBT-E) for eating disorders (Fairburn, 2008), without a mindfulness skills intervention
  Interventions: Behavioral: CBT-E

INTERVENTIONS:
Behavioral: MIND — Both experimental and control groups receive 20 weekly sessions (1.5 hours each), based on principles of CBT-E (Fairburn, 2008), adapted for a group format .
  The experimental group will receive in addition to CBT-E a mindfulness based intervention comprising of 4 weekly group sessions (1.5 hours each) during the month prior to the CBT-E program. The mindfulness skills intervention will also be practiced throughout the CBT-E program at the beginning of every group session and independently as homework. Mindfulness intervention includes "formal" mindfulness practice (brief mindfulness meditation - 10 minutes each) and "informal" mindfulness practice (Other "non meditation exercises", also known as "mindfulness in everyday life"- eg "STOP").
  Arms: Experimental group (CBTE-MIND)
Behavioral: CBT-E — The comparison group (control) will receive 4 weekly supportive-educational group sessions (1.5 hours each) prior to the group CBT-E program, with no mindfulness content or training.

SUMMARY:
Bulimia Nervosa (BN), Binge Eating Disorder (BED) and Night Eating Syndrome (NES) are Binge Eating Disorders (BE-Dis) in which binge eating episodes are a main symptom. Cognitive Behavioral Therapy (CBT) is the leading evidence-based treatment for patients suffering from these disorders. CBT-E is an "enhanced" trans-diagnostic version of the treatment which appears to be more effective in a variety of Eating Disorders (EDs). The main goals of this treatment are reducing dietary restrictions and EDs symptoms as well as food intake regulation. Self-monitoring (SM) is an important and central tool in this type of treatment considered crucial for its success. Therefore, during treatment, patients are required to monitor their eating, the circumstances, and their thoughts and feelings proximate to the time of eating. Nevertheless, despite the importance of this tool, research has shown that there are many difficulties challenging the clients' adherence to SM, which might reduce this treatment's effectiveness and outcome. Additionally, in recent years there has been cumulative data supporting the use of mindfulness in the treatment of EDs. Mindfulness, as a western psychological approach, is defined as the "unique non-judgmental focus of one's attention at the present moment". Although SM requires the ability to observe, describe and identify occurrences, no studies have yet examined the direct effect of mindfulness skills on SM adherence, and therefore the improvement of treatment outcomes.

The main objective of the present study is to examine the effect of a mindfulness based intervention on SM adherence during a CBT intervention for BE-Dis, and on the treatment outcomes as seen in the ED psychopathology and compliance to the nutritional instructions and food intake composition. Other aims include examining the differences between the experimental group and the control group, regarding their level of mindfulness and SM adherence. In addition, mediating and moderating processes between mindfulness and SM adherence will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 18-60 who meet the criteria for BN, BED or NES according to the DSM-V.
* The participants will be recruited via convenience sampling among patients applying for treatment in the ED unit in "Hanotrim" outpatient clinic ("Shalvata" mental health center) and through internet advertising.
* Participation in the research program will be allowed only after evaluation and a diagnostic procedure to examine if the criteria for CBT are met in terms of diagnosis and motivational status. This procedure will be conducted through psychological and nutritional intake.

Exclusion Criteria (contraindications to starting CBT-E immediately):

* Current suicidal ideation
* Current substance/alcohol dependence or abuse
* Current psychosis
* Pregnancy (which began prior inclusion)
* Inability to attend treatment on a regular basis

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2018-01-01 (Estimated); Study Completion 2018-01-01 (Estimated)

PRIMARY OUTCOMES:
Changes in the Eating Disorder Examination Questionnaire (EDE-Q-I) | 8 Time points: Recruitment (entry to study), pre-CBT-E (5 weeks from recruitment), along CBT-E (10, 5, 20 weeks from recruitment), post-CBT-E (24 weeks from recruitment), follow-up (3 and 6 months post CBT-E = 9 and 12 months post recruitment)
  EDE-Q-I (Eating Disorder Examination Questionnaire; Fairburn & Beglin, 1994): A self-report measure of eating disorders psychopathology.
Changes in the Clinical Impairment Assesment (CIA) questionnaire | 8 Time points: Recruitment (entry to study), pre-CBT-E (5 weeks from recruitment), along CBT-E (10, 5, 20 weeks from recruitment), post-CBT-E (24 weeks from recruitment), follow-up (3 and 6 months post CBT-E = 9 and 12 months post recruitment)
  Assessment of psychosocial impairment due to eating disorder will be conducted through CIA (Clinical Impairment Assesment) self-report questionnaire (Bohn & Fairburn, 2008).
Changes in the Night Eating Questionnaire (NEQ) | 8 Time points: Recruitment (entry to study), pre-CBT-E (5 weeks from recruitment), along CBT-E (10, 5, 20 weeks from recruitment), post-CBT-E (24 weeks from recruitment), follow-up (3 and 6 months post CBT-E = 9 and 12 months post recruitment)
  Assessment of Night Eating Syndrome psychopathology will be conducted through NEQ (Night Eating Questionnaire) self-report questionnaire (Allison et al., 2008).
Changes in the treatment Outcome Questionnaire-45 (OQ-45) | 8 Time points: Recruitment (entry to study), pre-CBT-E (5 weeks from recruitment), along CBT-E (10, 5, 20 weeks from recruitment), post-CBT-E (24 weeks from recruitment), follow-up (3 and 6 months post CBT-E = 9 and 12 months post recruitment)
  OQ-45 (Outcome Questionnaire-45) (Lambert et al., 1996) is a self-report scale used to estimate client degree of disturbance at the outset and over the course of treatment. It measures three subscales: symptom distress (depression and anxiety), interpersonal relationships and social role (difficulties in the workplace, school or home duties).
Treatment outcomes as seen in the compliance to the nutritional instructions (conducted through analyzing the self monitoring documents ) | Analyzed at 3 time points along the CBT-E program: week 1, week 10, week 19 (end of CBTprogram)
  Treatment outcomes regarding the compliance to the nutritional instructions, will be examined by analyzing the participants' self monitoring reports.
  This analysis will be conducted by comparing the actual number of meals a day and the composition of food consumed (and reported) to dietary recommendations for the treatment of binge eating disorders (Fairburn & Wilson, 1993).
  Nutritional composition analysis of food consumed will be conducted by using the "Tzameret" software (of the Israeli Ministry of Health).
  This procedure will be conducted before (week 1), during (week 10) and at the end of the CBT program (week 19).

SECONDARY OUTCOMES:
Self monitoring adherence (conducted through scoring the self monitoring content of the participants) | Every week along 19 weeks of CBTE program
  Self monitoring during the CBT-E program will be conducted electronically using the Qualtrics software via the participants' smartphones (for both groups).
  Adherence to self monitoring will be evaluated by analyzing and scoring the self monitoring content of each participant. In this procedure we are measuring every week along 19 weeks of CBTE program:
  * The number of days documented in the self monitoring form
  * The degree of detail type and quantity of food reported (The percentage of total reports)
  * The extent (frequency) of real-time monitoring (real-time monitoring will be examined by comparing the time gaps between the reported time of eating, and the actual electronic timestamp (The percentage of total reports)
  * The extent (frequency) which the participant used the thoughts\feelings column (The percentage of total reports)

OTHER OUTCOMES:
Mediating and moderating processes between mindfulness and SM adherence: Depression and anxiety (will be examined through self-report questionnaires) | 8 Time points: Recruitment (entry to study), pre-CBT-E (5 weeks from recruitment), along CBT-E (10, 5, 20 weeks from recruitment), post-CBT-E (24 weeks from recruitment), follow-up (3 and 6 months post CBT-E = 9 and 12 months post recruitment)
  Depression and anxiety: DASS-21 (Depression Anxiety Stress Scales-21) (Lovibond & Lovibond, 1995)
Mediating and moderating processes between mindfulness and SM adherence: Motivation (will be examined through self-report questionnaires) | 8 Time points: Recruitment (entry to study), pre-CBT-E (5 weeks from recruitment), along CBT-E (10, 5, 20 weeks from recruitment), post-CBT-E (24 weeks from recruitment), follow-up (3 and 6 months post CBT-E = 9 and 12 months post recruitment)
  Motivation: SCQ (Stages of Change Questionnaire) (McConnaughy, Prochaska, &Velicer, 1983)
Mediating and moderating processes between mindfulness and SM adherence: Attention deficit disorder (will be examined through self-report questionnaires) | 8 Time points: Recruitment (entry to study), pre-CBT-E (5 weeks from recruitment), along CBT-E (10, 5, 20 weeks from recruitment), post-CBT-E (24 weeks from recruitment), follow-up (3 and 6 months post CBT-E = 9 and 12 months post recruitment)
  Attention deficit disorder: ASRS (ADHD Self Report Scale) ( Kessler et al, 2005)
Mediating and moderating processes between mindfulness and SM adherence: Dissociation (will be examined through self-report questionnaires) | 8 Time points: Recruitment (entry to study), pre-CBT-E (5 weeks from recruitment), along CBT-E (10, 5, 20 weeks from recruitment), post-CBT-E (24 weeks from recruitment), follow-up (3 and 6 months post CBT-E = 9 and 12 months post recruitment)
  Dissociation: DES (Dissociative Experience Scale ) (Freyberger et al., 1998)
Mediating and moderating processes between mindfulness and SM adherence: Obsessiveness (will be examined through self-report questionnaires) | 8 Time points: Recruitment (entry to study), pre-CBT-E (5 weeks from recruitment), along CBT-E (10, 5, 20 weeks from recruitment), post-CBT-E (24 weeks from recruitment), follow-up (3 and 6 months post CBT-E = 9 and 12 months post recruitment)
  Obsessiveness: WISPI (Wisconsin Personality Disorder Inventory-4) (Klein et al., 1993)
Mediating and moderating processes between mindfulness and SM adherence: Impulsivity, perfectionism and interoceptive awareness (will be examined through self-report questionnaires) | 8 Time points: Recruitment (entry to study), pre-CBT-E (5 weeks from recruitment), along CBT-E (10, 5, 20 weeks from recruitment), post-CBT-E (24 weeks from recruitment), follow-up (3 and 6 months post CBT-E = 9 and 12 months post recruitment)
  Impulsivity, perfectionism and interoceptive awareness: EDI-2 (Eating Disorders Inventory-2) (Garner, 1991)
Mediating and moderating processes between mindfulness and SM adherence: therapeutic alliance (will be examined through self-report questionnaires) | 8 Time points: Recruitment (entry to study), pre-CBT-E (5 weeks from recruitment), along CBT-E (10, 5, 20 weeks from recruitment), post-CBT-E (24 weeks from recruitment), follow-up (3 and 6 months post CBT-E = 9 and 12 months post recruitment)
  Therapeutic alliance: WAI (Working Alliance Inventory)(Tracey & Kokotovic, 1989) - a self-report questionnaire.
Level of mindfulness | 8 Time points: Recruitment (entry to study), pre-CBT-E (5 weeks from recruitment), along CBT-E (10, 5, 20 weeks from recruitment), post-CBT-E (24 weeks from recruitment), follow-up (3 and 6 months post CBT-E = 9 and 12 months post recruitment)
  Assessment of changes in mindfulness levels throughout the treatment and the follow up period will be conducted via self-report questionnaire:
  FFMQ (Five Facet Mindfulness Questionnaire) (Baer, Smith, Hopkins, Krietemeyer & Toney, 2006)

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Steiner, MD, Study Director — Shalvata Mental Health Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fairburn, C. G. (2008). Cognitive behavior therapy and eating disorders. New York: Guilford Press